CLINICAL TRIAL: NCT05010304
Title: Penicillin De-labeling in the Pediatric Primary Care Setting
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: American College of Allergy, Asthma and Immunology (Other)
Responsible Party: Principal Investigator, Timothy Chow, MD, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STU-2021-0517
Record Dates: First submitted 2021-08-10; First posted 2021-08-18 (Actual); Results first posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-07

CONDITIONS: Penicillin Allergy; Penicillin Reaction
Keywords: penicillin; allergy
MeSH Terms: conditions — Hypersensitivity | interventions — Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pediatric Patients with a history of penicillin allergy (Experimental)
  Interventions: Drug: Amoxicillin

INTERVENTIONS:
Drug: Amoxicillin — Two-dose amoxicillin challenge

SUMMARY:
While reported adverse reactions to penicillins are common, most patients with a penicillin allergy label can safely tolerate penicillins, and elective evaluation for penicillin allergy has been recommended. For low-risk patients, direct oral challenge may be an optimal approach as a delabeling strategy. However, there is a vast disparity between the number of patients with a penicillin allergy label and practicing allergists in the United States, and implementing outpatient primary care-based delabeling strategies in low-risk patients may increase access to delabeling assessments. However, a recent survey of pediatricians identified perceived barriers to implementing penicillin allergy evaluations into their routine care. Significant gaps in knowledge exist regarding the feasibility of this approach involving risk stratification evaluation of reported penicillin adverse reactions and direct amoxicillin challenge procedures in low-risk patients in the pediatric primary care setting. With this, the primary aim of this study is to evaluate the number of patients for which risk-stratification and direct amoxicillin challenge are successfully completed in an outpatient pediatric primary care clinic.

ELIGIBILITY:
Inclusion Criteria:

* Children from ages 2-18 years with a history of parent-reported penicillin allergy.

Exclusion Criteria:

* Children with a history of reaction consistent with a severe cutaneous adverse reaction to penicillin as defined as a history of oral blisters, diffuse skin peeling or blisters after taking a penicillin, or having the diagnosis of Stevens Johnson Syndrome, Toxic Epidermal Necrolysis, Drug rash with eosinophilia and systemic symptoms will be excluded. Pregnant and breastfeeding female subjects will be excluded

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-11-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Medical Center Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chow TG, Patel G, Mohammed M, Johnson D, Khan DA. Delabeling penicillin allergy in a pediatric primary care clinic. Ann Allergy Asthma Immunol. 2023 May;130(5):667-669. doi: 10.1016/j.anai.2023.01.034. Epub 2023 Feb 2. No abstract available. PMID 36738783

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pediatric Patients With a History of Penicillin Allergy
Started | 23
Completed | 23
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pediatric Patients With a History of Penicillin Allergy
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.3 (0.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Subjects Who Complete Risk-stratification of Penicillin Allergy in the Pediatric Primary Care Setting
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Pediatric Patients With a History of Penicillin Allergy
Number analyzed (Participants) | 23
Participants | 23

2. Primary Outcome: Subjects Stratified as Low-risk With a Negative Immediate Amoxicillin Challenge in the Pediatric Primary Care Setting
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Pediatric Patients With a History of Penicillin Allergy
Number analyzed (Participants) | 23
Participants | 21

3. Secondary Outcome: Penicillin Allergy Labeling in Subjects With Negative Amoxicillin Challenge
Description: Subjects who have a penicillin allergy label added back to their electronic health record at 10-14 months after amoxicillin challenge.
Time Frame: 10-14 months after amoxicillin challenge
Measure: Count of Participants; unit: Participants
Arm/Group | Pediatric Patients With a History of Penicillin Allergy
Number analyzed (Participants) | 21
Participants | 0

ADVERSE EVENTS:
Time Frame: 7 days after amoxicillin challenge completion
Description: Adverse events were captured by study staff during the 60 minute observation period with amoxicillin challenge, and again assessed at 7 days after challenge completion by study staff.
Arm/Group | Pediatric Patients With a History of Penicillin Allergy
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 2/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pediatric Patients With a History of Penicillin Allergy (N=23)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) — Cutaneous-only reaction, resolving with oral antihistamines

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-29): https://cdn.clinicaltrials.gov/large-docs/04/NCT05010304/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-06): https://cdn.clinicaltrials.gov/large-docs/04/NCT05010304/ICF_001.pdf